CLINICAL TRIAL: NCT06449573
Title: Evaluation of Cardiopulmonary Parameters in Individuals With Asthma
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aydan Aslı Aksel Uylar, Physiotherapist, Hacettepe University
Other Study IDs: GO 23/533
Record Dates: First submitted 2024-03-03; First posted 2024-06-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: Inclusion Criteria:
  * Patients receiving step 5 asthma treatment
  * 18-65 years
  * Asthma under control (asthma control test ≥20)
  * No more than 2 exacerbations in the last 1 year
  Exclusion Criteria:
  * Non-consenting
  * Patients with asthma exacerbation requiring systemic steroid use for at least 3 days in the last 1 month
  * Being an active smoker
  Interventions: Other: Exercise capacity
- Healthy Individuals: Inclusion Criteria:
  * No respiratory, cardiovascular and metabolic diseases
  * Regular non-smoker
  Exclusion Criteria:
  * Non-consenting
  * Pregnant women
  Interventions: Other: Exercise capacity

INTERVENTIONS:
Other: Exercise capacity — cardiopulmonary exercise test used assessment of exercise capacity

SUMMARY:
The aim of the study compare the cardiopulmonary parameters of individuals with asthma with healthy subjects.

DETAILED DESCRIPTION:
It is thought that aerobic capacity of asthmatic individuals decreases due to chronic respiratory disease, especially oxygen consumption. Detailed investigation will be provided with this research.

ELIGIBILITY:
Inclusion Criteria:

* No respiratory, cardiovascular and metabolic diseases
* Regular non-smoker

Exclusion Criteria:

* Non-consenting
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include asthma patients followed up by Hacettepe University Faculty of Medicine, Department of Chest Diseases, Immunology and Allergy Branch and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 20 minutes
  Exercise capacity will be assessed by Cardiopulmonary Exercise Test. The test will be performed on a bicycle ergometer. The test will be terminated when the target heart rate is reached or when the patient indicates that they are unable to continue the test. maximal oxygen consumption and the workload achieved will be recorded.

SECONDARY OUTCOMES:
Respiratory muscle strength | 8 minutes
  Inspiratory and expiratory muscle strength will be measured with a mouth pressure measuring device. Measurements will be made in a sitting position with the hip and knee at 90 degrees and the trunk upright.
Peripheral muscle strength | 5 minutes
  It will be evaluated with a portable manual muscle strength measuring device. Muscle strength of knee extensors will be measured. The measurement will be performed with the patient sitting with his/her back unsupported and his/her hands crossed on his/her chest.
Grip strength | 3 minutes
  It will be evaluated with a portable hand dynamometer. Measurements will be made in a sitting position with the hip and knee at 90 degrees and the trunk upright. The measurement will be performed with the arm adjacent to the side of the trunk and the forearm parallel to the ground.
Kinesiophobia | 3 minutes
  Tampa Kinesiophobia Scale will be used. A total of 17 questions will be answered in 4-point Likert form. In total, the patient scores between 17-68. A high score indicates high kinesiophobia.
Quality of Life (symptoms, mood, activity limitation, environmental exposure) | 10 minutes
  Asthma Quality of Life Scale will be used for the evaluation. This scale consists of 4 sub-headings including symptoms, mood, activity limitation, environmental exposure and 32 questions. Each item is scored between 1-7. The total score of the scale is calculated by averaging the scores given to the items. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar Yagli, Study Director — Hacettepe University; Melda Saglam, Study Chair — Hacettepe University; Ebru Damadoglu, Study Chair — Hacettepe University; Merve Firat, Study Chair — Kirsehir Ahi Evran Universitesi; Aydan Aslı Aksel Uylar, Principal Investigator — Hacettepe University; Melek Cihanbeylerden, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)